CLINICAL TRIAL: NCT00210431
Title: A Post Marketing Surveillance Study of Dysport Formulated With a Batch of Bulk Active Substance From a New Primary Manufacturing Facility at the Centre for Applied Microbiology & Research (CAMR)
Brief Title: Post Marketing Surveillance Study of Dysport
Status: Completed | Type: Observational
Sponsor: Ipsen (Industry)
Other Study IDs: Y-47-52120-093
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Blepharospasm; Hemifacial Spasm; Cervical Dystonia; Spasmodic Torticollis; Cerebral Palsy; Muscle Spasticity; Cerebrovascular Accident; Equinus Deformity; Facial Hyperdynamic Lines
MeSH Terms: conditions — Blepharospasm; Hemifacial Spasm; Torticollis; Cerebral Palsy; Muscle Spasticity; Stroke; Equinus Deformity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

SUMMARY:
The purpose of this study is to provide further information regarding the risks and benefits of Dysport in marketed indications.

ELIGIBILITY:
Inclusion Criteria:

* adult or child over the age of 2 years
* scheduled to receive Dysport as per their normal treatment practice, and in conformance with their country's Summary of Product Characteristics

Exclusion Criteria:

* history of hypersensitivity to Dysport or drugs with a similar chemical structure
* treatment with any other investigational drug within the last 30 days before survey entry

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 783 (Actual)
Dates: Start 2004-10; Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
- assessment of efficacy as assessed by treating physician at scheduled follow up visit
- data on adverse events since treatment with Dysport

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (36):
- France (17):
  - Centre Hospitalier Saint Esprit, Agen
  - Center Hospitalier du Pays d'Aix, Aix-en-Provence
  - Centre Hospitalier, Chambéry
  - Hopital Timone Adultes, Marseille
  - Hopital Central, Nancy
  - Hopital Hotel Dieu, Nantes
  - Hopital Pasteur, Nice
  - Hopital Caremeau, Nîmes
  - Hopital Saint Antione, Paris
  - Centre Hospitalier Pitie Salpetriere, Paris
  - Hopital Sainte Anne, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - CHU Charles Nicolle, Rouen
  - Hopital Bellevue, Saint-Etienne
  - Hopital Civil, Strasbourg
  - Hopital Purpan, Toulouse
  - Hopital Rangueil, Toulouse
- Germany (9):
  - Praxis für Neurologie, Berlin
  - Rhein. F.-Wilhelms-Universität, Bonn
  - Praxis für Neurologie, Giessen
  - Städt. Krankenhaus Martha-Maria, Halle-Dölau
  - Neurologische Praxis, Hamburg
  - Med. Hochschule, Hanover
  - Bürgerhospital, Stuttgart
  - E.-Karls-Universität, Tübingen
  - Klinikum der Stadt Villingen-Schwenningen, Villingen-Schwenningen
- Russia (10):
  - Alma-Ata State Institute of Postgraduate Education, Alma-Ata, Kazakhstan
  - Rehabilitation Centre "Balbulak", Alma-Ata, Kazakhstan
  - Centre of plastic surgery "Reconstruction and Recreation", Moscow
  - Institute of Medical Aestetic "Vallex-M", Moscow
  - Moscow Medical Academy, Moscow
  - Scientific Research Institute of Neurology, Moscow
  - Cosmetological Centre "Diamond", Moscow
  - National Medical Centre of Surgery, Moscow
  - Federal Centre "Pediatric Rehabilitology", Moscow
  - Centre for Aesthetic Dermatology and Surgery of Russian Academy of Sciences, Moscow